CLINICAL TRIAL: NCT04422574
Title: COVID 19 Serology in Pulmonologists : Pneumo Sero Cov
Brief Title: COVID 19 Serology in Pulmonologists
Acronym: Pneumoserocov
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0343
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Covid 19
Keywords: Covid 19; serology
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Respiratory physicians are highly exposed workers to Covid-19 as they perform spirometry, endoscopy, and manage Covid-19 in first line for most of them. Moreover, none reported to have apply increased levels of protection for performing these acts in the most active period of viral circulation, until the lockdown. Whether they were most frequently immunized against SARS-CoV-2 at the end of the first wave than the general population is of utmost importance individually but also worldwide

ELIGIBILITY:
Inclusion Criteria:

* Pulmonologists of Languedoc Roussillon
* Actively working
* Registered

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonologists of Languedoc Roussillon
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
covid 19 serology | 1 day
  covid 19 serology with cross sectional
risk factors for positive serology testing | 1 day
  risk factors for positive serology testing with cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC